CLINICAL TRIAL: NCT00875082
Title: Effect of Montelukast on Metalloproteinase (MMP)-9, MMP-12, Tissue Inhibitor Metalloproteinase-1 (TIMP-1), Procollagen Type I C-terminal Peptide (PICP) and TGF-beta1 Levels in Sputum From Mild Intermittent Asthmatic Children: a Pilot Study
Brief Title: Effect of Montelukast on Remodelling Markers in Asthmatic Children
Acronym: MORACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Boner Attilio, Prof, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UVAB-02
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Asthma; Children; Remodelling; Metalloproteinases; Montelukast
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): Montelukast chewing tablets once daily per os, plus inhaled short acting beta2 agonist as needed
  Interventions: Drug: Montelukast
- placebo (Placebo Comparator): placebo chewing tablets per os once daily, plus inhaled short acting beta 2 agonist as needed
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast, chewing tablets 5mg, once daily, 8 weeks
  Arms: Montelukast
Drug: placebo — placebo chewing tablets once daily, plus inhaled short acting beta2 agonist as needed, 8 weeks
  Arms: placebo

SUMMARY:
Airway smooth muscle cell layer thickening and sub epithelial fibrosis, key allergen-induced airway remodelling features not modulated by corticosteroids, are reversible by CysLT1 receptor blockade therapy in animals. No data are available, at the present, about the potential effect of LTs receptor antagonists on airway remodelling in asthmatic children.

In the present study, the investigators aim to assess whether the addition of montelukast to ICS in mild asthmatic children to inhibit the release of MMP-9, TIMP-1, MMP-12, MMP-9/TIMP1 ratio, procollagen type I C-terminal peptide (PICP) and TGF-beta in the airway fluid collected by induced sputum in asthmatic children. 30-40 atopic children with mild persistent asthma.

Children with asthma will be recruited and evaluated with a real life open label trial: they will be randomised into two groups at first visit (T1): 1) group A: in these patients montelukast tablets 5 mg and as needed beta agonist will be administered; 2) group B: in these patients beta agonist therapy only.

All children will be evaluated after 8 weeks (T2). They will be tested for lung function, FeNO, metalloproteinase (MMP)-9, MMP-12, tissue inhibitor metalloproteinase-1 (TIMP-1), procollagen type I C-terminal peptide (PICP) and TGF-beta1 levels in sputum.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria: the classification of asthma will be based on clinical history and examination and pulmonary function parameters, according to international guidelines.
* Stage and/or severity of condition: atopic children with mild intermittent asthma will be enrolled. Atopy will be evaluated by skin-prick test to common allergens in the area.
* Confirmatory physical and laboratory findings:
* Age: ranging in age 6 to 14 years.
* Evidence of susceptibility to the disease under study
* Patients have not used ICS during 3-month period prior to study entry

Exclusion Criteria:

* Patients will be excluded if they had used oral steroids in the last month.
* Patients will be excluded if they had acute or chronic lung diseases other than asthma, upper or lower airway infection in the previous 3 weeks or during the trial, acute asthma exacerbation, or had used oral steroids in the last month.
* Patients will be excluded if they had acute or chronic lung diseases other than asthma, upper or lower airway infections in the previous 3 weeks or during the trial, acute asthma exacerbation, or had used oral steroids in the last month.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
FeNo, Lung Function, MMP-9, MMP-12, TIMP-1, PICP and TGFB determination | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Attilio L Boner, MD, Principal Investigator — Pediatric Department, Università di Verona
Locations (1):
- Pediatric Department, University of Verona, Verona, Italy

REFERENCES:
- [Derived] Tenero L, Piazza M, Sandri M, Azzali A, Chinellato I, Peroni D, Boner A, Piacentini G. Effect of montelukast on markers of airway remodeling in children with asthma. Allergy Asthma Proc. 2016 Sep;37(5):77-83. doi: 10.2500/aap.2016.37.3978. PMID 27657514